CLINICAL TRIAL: NCT01831115
Title: Basics in Acute Shortness of Breath EvaLuation (BASEL V) Study
Acronym: BASEL V
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: BASEL V
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dyspnea
Keywords: heart failure; BNP; acute dyspnoea
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA, Plasma and Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
To improve the diagnostic and prognostic utility of various biomarkers, detailed patient's history, physical examinations and technical devices in patients presenting with acute dyspnea.

DETAILED DESCRIPTION:
Background: Acute heart failure is a common disease associated with high morbidity and mortality. Unfortunately, pathophysiology and optimal initial treatment are both ill defined.

Working Hypothesis:

* Improved understanding of the pathophysiology underlying heart failure might allow more cause-specific treatment to this syndrome.
* More rapid diagnosis of acute heart failure may allow to more rapidly initiate the appropriate treatment.
* Cardiac dysfunction especially in comorbid dyspneic patients is not adequately characterized and the spectrum of acute heart failure is more diverse than originally thought.

Methods: This is a large multicenter center, observational study enrolling unselected, consecutive patients with acute dyspnea presenting to the Emergency Department. Patient history, physical examination and laboratory parameters will be systematically obtained. Echocardiographic examinations will be routinely performed. Follow-up will be done at specified intervals (3, 6 and 12 months) after the initial presentation and risk predictors will be analyzed in multivariable regression models.

Expected Value of the Proposed Project: The data obtained during this project will help to further improve diagnostics and prognostics in patients with acute dyspnea and to better understand underlying pathology of cardiac dysfunction in this cohort.

Significance: The study aims are up-to-date and deal with an important health care problem in society. Conclusions drawn will significantly change care of patients with acute heart failure probably leading to a significant reduction of rehospitalization, morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* chief complaint of dyspnea (not penetrating injury or trauma related)
* subjects must be at least 18 years of age

Exclusion Criteria:

* patient is unable or unwilling to give informed consent
* patient on hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute dyspnea to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 5452 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for the diagnosis of heart failure | baseline
  Diagnostic of various biomarkers (such as natriuretic peptides, cardiac troponins, microRNA...), physical examination, detailed patient's history and novel technical devices.
Prognostic utility in patients with dyspnea | 360 days
  Prognostic value of various biomarkers, echocardiography data and novel technical measurements regarding rehospitalisation, cardiovascular mortality and all-cause and mortality
Prognostic utility in patients with dyspnea | 720 days
  Prognostic value of various biomarkers, echocardiography data and novel technical measurements regarding rehospitalisation, cardiovascular mortality and all-cause and mortality

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zurich, Zurich

REFERENCES:
- [Derived] Belkin M, Wussler DN, Shrestha S, Lopez-Ayala P, Nowak A, Michou E, Papachristou A, Popescu C, Strebel I, Kozhuharov N, Sabti Z, Netzer I, Zimmermann T, Diebold M, Breidthardt T, Mueller C. Prognostic value of health-related quality of life in patients with acute dyspnoea: a cohort study. Swiss Med Wkly. 2025 Apr 15;155:3785. doi: 10.57187/s.3785. PMID 40450733
- [Derived] Belkin M, Wussler D, Michou E, Strebel I, Kozhuharov N, Sabti Z, Nowak A, Shrestha S, Lopez-Ayala P, Prepoudis A, Stefanelli S, Schafer I, Mork C, Albus M, Danier I, Simmen C, Zimmermann T, Diebold M, Breidthardt T, Mueller C. Prognostic Value of Self-Reported Subjective Exercise Capacity in Patients With Acute Dyspnea. JACC Adv. 2023 May 26;2(3):100342. doi: 10.1016/j.jacadv.2023.100342. eCollection 2023 May. PMID 38939580
- [Derived] Breidthardt T, van Doorn WPTM, van der Linden N, Diebold M, Wussler D, Danier I, Zimmermann T, Shrestha S, Kozhuharov N, Belkin M, Porta C, Strebel I, Michou E, Gualandro DM, Nowak A, Meex SJR, Mueller C. Diurnal Variations in Natriuretic Peptide Levels: Clinical Implications for the Diagnosis of Acute Heart Failure. Circ Heart Fail. 2022 Jun;15(6):e009165. doi: 10.1161/CIRCHEARTFAILURE.121.009165. Epub 2022 Jun 7. PMID 35670217
- [Derived] Diebold M, Kozhuharov N, Wussler D, Strebel I, Sabti Z, Flores D, Shrestha S, Martin J, Staub D, Venge P, Mueller C, Breidthardt T. Mortality and pathophysiology of acute kidney injury according to time of occurrence in acute heart failure. ESC Heart Fail. 2020 Oct;7(5):3219-3224. doi: 10.1002/ehf2.12788. Epub 2020 Jun 24. PMID 32578962
- [Derived] Wussler D, Kozhuharov N, Tavares Oliveira M, Bossa A, Sabti Z, Nowak A, Murray K, du Fay de Lavallaz J, Badertscher P, Twerenbold R, Shrestha S, Flores D, Nestelberger T, Walter J, Boeddinghaus J, Zimmermann T, Koechlin L, von Eckardstein A, Breidthardt T, Mueller C. Clinical Utility of Procalcitonin in the Diagnosis of Pneumonia. Clin Chem. 2019 Dec;65(12):1532-1542. doi: 10.1373/clinchem.2019.306787. Epub 2019 Oct 15. PMID 31615771
- [Derived] Wussler D, Kozhuharov N, Sabti Z, Walter J, Strebel I, Scholl L, Miro O, Rossello X, Martin-Sanchez FJ, Pocock SJ, Nowak A, Badertscher P, Twerenbold R, Wildi K, Puelacher C, du Fay de Lavallaz J, Shrestha S, Strauch O, Flores D, Nestelberger T, Boeddinghaus J, Schumacher C, Goudev A, Pfister O, Breidthardt T, Mueller C. External Validation of the MEESSI Acute Heart Failure Risk Score: A Cohort Study. Ann Intern Med. 2019 Feb 19;170(4):248-256. doi: 10.7326/M18-1967. Epub 2019 Jan 29. PMID 30690646
- [Derived] Badertscher P, Strebel I, Honegger U, Schaerli N, Mueller D, Puelacher C, Wagener M, Abacherli R, Walter J, Sabti Z, Sazgary L, Marbot S, du Fay de Lavallaz J, Twerenbold R, Boeddinghaus J, Nestelberger T, Kozhuharov N, Breidthardt T, Shrestha S, Flores D, Schumacher C, Wild D, Osswald S, Zellweger MJ, Mueller C, Reichlin T. Automatically computed ECG algorithm for the quantification of myocardial scar and the prediction of mortality. Clin Res Cardiol. 2018 Sep;107(9):824-835. doi: 10.1007/s00392-018-1253-z. Epub 2018 Apr 17. PMID 29667014
- [Derived] Breidthardt T, Moreno-Weidmann Z, Uthoff H, Sabti Z, Aeppli S, Puelacher C, Stallone F, Twerenbold R, Wildi K, Kozhuharov N, Wussler D, Flores D, Shrestha S, Badertscher P, Boeddinghaus J, Nestelberger T, Gimenez MR, Staub D, Aschwanden M, Lohrmann J, Pfister O, Osswald S, Mueller C. How accurate is clinical assessment of neck veins in the estimation of central venous pressure in acute heart failure? Insights from a prospective study. Eur J Heart Fail. 2018 Jul;20(7):1160-1162. doi: 10.1002/ejhf.1111. Epub 2018 Jan 4. No abstract available. PMID 29314487